CLINICAL TRIAL: NCT07219901
Title: Early Intervention in Infants With Unrepaired Cleft Palate: Language, Palatal Function, and Articulation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Old Dominion University (Other)
Collaborators: Children's Hospital of The King's Daughters (Other)
Responsible Party: Principal Investigator, Victoria Reynolds, Assistant Professor, Old Dominion University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2355082-5
Record Dates: First submitted 2025-10-16; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Cleft Lip and Cleft Palate; Cleft Lip Palate; Cleft Lip and/or Palate; Cleft Palate; Cleft Palate Children; Cleft Palates; Cleft Palate Repair
Keywords: cleft-type speech; hypernasality; palatal function; compensatory speech patterns; obligatory speech patterns; velopharyngeal dysfunction; communication; language; speech
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Communication; Language; Speech | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All participants will be allocated to this arm; they will receive the intervention as detailed elsewhere in this protocol.
  Interventions: Behavioral: Early intervention for language, articulation and palatal function skills

INTERVENTIONS:
Behavioral: Early intervention for language, articulation and palatal function skills — This intervention will use the principles of focused stimulation, and enhanced milieu teaching, to coach families in the following speech and language development strategies: attempting oral plosives, increasing phonetic inventory, mapping words to gesture use, and promoting canonical babbling.

SUMMARY:
The goal of this clinical trial is to learn if teaching speech skills to infants with cleft palates, prior to palate repair, will help them to develop speech and language skills. It will also learn about whether the skills are linked to fewer speech sound difficulties when they start school. The main questions it aims to answer are:

Do standard, early intervention techniques to promote language development, that are used in children who are late talkers, work in infants with cleft palates? Will infants with cleft palates increase the number of sounds they use after targeted intervention? Can infants attempt to make stop sounds, like b and p, after targeted intervention? Can infants with cleft palate learn new words more quickly when they are used with gestures?

Participants will:

Participate in a baseline evaluation of speech and language skills, either in person, or via Telehealth.

Attend the clinic for twice-weekly visits, for six weeks, to learn techniques to help their infants develop their speech and language skills, in a group setting with other families of infants with cleft palate.

Participate in a final evaluation of speech and language skills, either in person, or via Telehealth.

DETAILED DESCRIPTION:
Participants

Participants will be caregiver-infant dyads, where the infant is aged between six and twelve months at the time of study enrolment. Infants should be under the current care of a craniofacial team, with no medical diagnosis that would preclude study participation (e.g., reliance on supplementary oxygen, nasopharyngeal airway in situ).

Caregivers

Caregivers should be over the age of 18 years at the time of study enrolment and be able to participate in the group intervention in the English language, although they may speak more than one language or dialect. Individuals who are not able to consent to study participation (due to the presence of a health condition impeding the ability to give consent) will be excluded from this study. Caregivers should identify either as a primary, or joint-primary, caregiver for the infant. Individuals who are not primary caregivers, but who spent a significant amount of time with the infant and who interact with the infant, are also eligible for study participation. There is no limit on the number of caregivers who can attend sessions with their child, to account for non-traditional family structures.

Recruitment

Recruitment will take place at the Cleft and Craniofacial Center of the Children's Hospital of the King's Daughters. Recruitment flyers will be posted in the clinic (see attached recruitment flyer). Families will be invited to participate in the study no more than three times: once between birth and three months of age, at a cleft team meeting; once between three and six months of age at a cleft team meeting, and once again at the six to nine month visit (see attached recruitment script). Families will be invited a maximum of three times, or until first refusal, whichever comes first.

Caregivers will be provided with an information sheet about the study and two consent forms; one for their participation and one for their child's participation. These will be provided by the Surgical Services Unit Research Coordinator (SSURC), at clinic visits. Families will be asked if they would like more information about the study and given a verbal overview of the study and its participation requirements. The SSURC will then leave the clinic room for a brief period to give families time to read the consent forms. On her return, she will ask families if they have any questions, respond to these, and consent families formally, if they are agreeable.

Initial and final evaluations

In order to describe and understand the clinical population, caregivers will be asked to complete the MacArthur-Bates Communicative Development Inventory (MBCDI), which is a measure of understanding and use of words and gestures to communicate, in infants and toddlers aged up to 18 months. This will be the primary, language outcome measure. Additionally, the Rossetti Infant-Toddler Development Scale (RITDS) will be administered by the speech-language pathologist, cooperatively with the caregiver, to describe and understand aspects of communication beyond receptive and expressive language (e.g., pragmatics, attachment). As part of these evaluation sessions, a ten-minute interaction between the infant and the caregiver will be recorded, and a count of communicative behaviors (as outlined in the data sheet) will be made, after the end of the session.

Intervention protocol

The intervention will be delivered face-to-face, in a room in the Lions Child Study Center at Old Dominion University (205). Twelve sessions are planned, with two sessions per week over six weeks; a different topic area, and associated targets, will be selected and focused on each week.

An example, weekly session plans from the intervention protocol are included as an Appendix to this document. It is anticipated that sessions will last for one-hour, and by led by one or more licensed and credentialled speech-language pathologists. The corresponding home carryover handouts are also provided.

Experimental design

This pilot study will be a quasi-experimental, repeated-measures design, where participants serve as their own controls. Baseline data on each outcome measure will be collected at the initial evaluation, prior to commencement of the program, and again at the first group session. Families will be provided with questionnaire measures prior to the appointment, and ten minutes of caregiver-child interactions will be videorecorded for later analysis of outcomes that are measured by behavioral counts. Following the program, an individual, final evaluation and de-brief will be conducted where post-intervention data will be collected. Post-intervention data will be compared against pre-intervention data.

Statistical analysis

Pre- and post-intervention scores will be compared. Statistical test selection will depend on data distribution; although, as this pilot study is anticipated to have a small sample size, it is hypothesized that data will not be distributed normally, thus necessitating the use of non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Infants with unrepaired cleft palate (with or without cleft lip)
* Aged between 6 and 10 months at the time of study commencement

Exclusion Criteria:

* Medically fragile status that would preclude participation in this community-based study.
* Palatoplasty completed.
* Aged over one year
* Infants with cleft lip only

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-10-21 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
MBCDI (W&G) | From enrollment to the end of treatment at 8 weeks.
  Number of words and concepts, as measured by the MacArthur-Bates Communicative Development Inventory (Words and Gestures)

SECONDARY OUTCOMES:
Plosive attempts | From enrollment until the end of treatment at 8 weeks.
  Attempts at oral plosive phonemes
Phonemes | From enrollment to the end of treatment at 8 weeks.
  Number of different phonemes spontaneously produced by the infant.
Canonical babbling: frequency | From enrollment to the end of treatment at 8 weeks.
  Frequency of canonical babbling will be measured by counting the number of canonical babblings produced by the infant in a ten-minute, caregiver-infant interaction.
Canonical babbling: shape | From enrollment to the end of treatment at 8 weeks.
  Shape of canonical babbling will be measured by recording and phonotactically transcribing the syllable shapes of canonical babbling observed during a ten-minute caregiver-infant interaction. The number of different shapes will be calculated.
Words versus gestures | From study enrollment to end of treatment at 8 weeks.
  Number of words, protowords and/or word attempts, relative to the number of communicative gestures produced.

OTHER OUTCOMES:
Caregiver confidence | From enrollment to end of treatment at 8 weeks.
  Each Q will be rated on a scale of 0 - 10: 0 = complete absence, 10 = full confidence. The total score will be calculated from the sum of scores for each question.
  How confident are you:
  Practicing language development strategies with your child? Knowing how your child should be playing for their age? Engaging in communication with your child (e.g., face-to-face, playing with a ball)? Taking turns with your child, in conversation (e.g., baby makes a sound, you repeat the sound) and play (e.g., you roll the ball, they roll the ball)? Knowing how your child should be babbling for their age? Knowing which sounds are impacted by having a cleft palate? Redirecting your child when they use throat sounds? Interpreting your child's gestures? Connecting their gestures to their/your spoken words? Promoting lip and tongue movements in your child? Helping your child to make new sounds? Overall, in supporting your child's speech and language development?
Conversational turn-taking: length of conversational utterance | From enrollment to end of treatment at 8 weeks
  Increase the length of conversational turn-taking in infant-caregiver interactions. Conversational turns, within a ten minute period, will be measured with a stopwatch. This value (length) will be calculated from the mean (or median, depending on data distribution) duration of the caregiver's conversational turn, in seconds.
Conversational turn-taking: frequency of conversational utterance | From enrollment to end of treatment at 8 weeks
  Increase the frequency of conversational turn-taking in infant-caregiver interactions. Conversational turns, within a ten minute period, will be counted. The total number of conversational turns will be used as the outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Reynolds, LLB BSc PhD, Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
We do not believe that we have Institutional Review Board (IRB) approval for this level of data sharing.